CLINICAL TRIAL: NCT00518089
Title: A Study of the Safety and Efficacy of Gatifloxacin in Patients With Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 198782-005
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Gatifloxacin; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Gatifloxacin 0.5% Eye Drops (Experimental): Gatifloxacin 0.5% Eye Drops
  Interventions: Drug: Gatifloxacin 0.5% eye drops
- Placebo Eye Drops (Placebo Comparator): Placebo Eye Drops
  Interventions: Drug: placebo eye drops

INTERVENTIONS:
Drug: Gatifloxacin 0.5% eye drops — Day 1 = 1 drop of study medication every 2hrs up to 8 times total; day 2-5 = 1 drop twice daily
  Arms: Gatifloxacin 0.5% Eye Drops
Drug: placebo eye drops — Day 1 = 1 drop of study medication every 2hrs up to 8 times total; day 2-5 = 1 drop twice daily
  Arms: Placebo Eye Drops

SUMMARY:
The study will determine the safety and efficacy of gatifloxacin eye drops in patients with bacterial conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with bacterial conjunctivitis

Exclusion Criteria:

* Signs and/or symptoms of conjunctivitis for more than 96 hours
* Signs and/or symptoms suggestive of fungal, viral, or allergic conjunctivitis
* Clinical diagnosis of chlamydia in either eye

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Downey, California, United States
- RajajiNagar, Bangalore, India

REFERENCES:
- [Background] Heller W, Cruz M, Bhagat YR, De Leon JM, Felix C, Villanueva L, Hollander DA, Jensen H. Gatifloxacin 0.5% administered twice daily for the treatment of acute bacterial conjunctivitis in patients one year of age or older. J Ocul Pharmacol Ther. 2014 Dec;30(10):815-22. doi: 10.1089/jop.2014.0040. PMID 25244402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Started | 430 | 429
Completed | 402 | 398
Not Completed | 28 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops | Total
Number analyzed (Participants) | 430 | 429 | 859
Age, Customized [Number; unit: participants]
  1-18 years | 66 | 74 | 140
  19-65 years | 316 | 313 | 629
  >65 years | 48 | 42 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 156 | 339
  Male | 247 | 273 | 520

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Patients With Clearing (Clinical Success) of Conjunctival Hyperemia and Conjunctival Discharge at Day 6
Description: Percentage of patients that achieved clinical success, defined as achievement of a score of zero for both conjunctival hyperemia and conjunctival discharge in the study eye at Day 6. Conjunctival hyperemia and conjunctival discharge were each assessed on a 4-point severity grade scale (0=none, +1=mild, +2=moderate, +3=severe).
Time Frame: Day 6
Population: Modified Intent to Treat; defined as all randomized patients who were "culture positive" at baseline meaning the culture of the eye grew bacteria. (Note: The Day 6 analysis included all Day 6 visit data, regardless of whether it was collected on Day 6 or on a later day).
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 166 | 167
Percentage of Patients | 59.6 | 46.7

2. Secondary Outcome: Percentage of Patients With Microbiological Cure Up to Day 6
Description: Percentage of patients with microbiological cure, defined such that all bacteria present in the study eye at Day 1 (Baseline) are eradicated up to Day 6 based on a Classification of Microbial Response. (Eradication=pathogen is absent in follow-up culture; Reduction=pathogen is reduced from baseline below threshold count in follow-up culture; Persistence=pathogen reduced from baseline but is above or equal to threshold count in follow-up culture; and Proliferation=pathogen has increased in count from baseline in follow-up culture).
Time Frame: 6 Days
Population: Modified Intent to Treat; defined as all randomized patients who were "culture positive" at baseline meaning the culture of the eye grew bacteria. (Note: The "Up to Day 6" analysis included all data up to the Day 6 time point but excluded any Day 6 visit data that was collected after the Day 6 time point).
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 166 | 167
Percentage of Patients | 92.2 | 80.2

3. Secondary Outcome: Percentage of Patients With Clinical Improvement of Ocular Signs Up to Day 6
Description: Percentage of patients with clinical improvement of ocular signs up to Day 6 based on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe), defined as a decrease (improvement) from Day 1 (Baseline) in the total score of conjunctival hyperemia and mucopurulent discharge (pus), with no increase (worsening) from Day 1 (Baseline) in either individual variable in the study eye.
Time Frame: 6 Days
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 166 | 167
Percentage of Patients | 97.0 | 92.2

4. Secondary Outcome: Percentage of Patients With Clinical Improvement of Ocular Symptoms Up to Day 6
Description: Percentage of patients with clinical improvement of ocular symptoms, defined as a decrease (improvement) up to Day 6 from Day 1 (Baseline) in the total score of itching and tearing (each on 4-point scale: 0 = none, 1 = mild, 2 = moderate, and 3 = severe), with no increase (worsening) from Day 1 (Baseline) in any individual score in the study eye diagnosed with bacterial conjunctivitis.
Time Frame: 6 Days
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 166 | 167
Percentage of Patients | 92.8 | 88.6

5. Primary Outcome: Percentage of Patients With Clearing (Clinical Success) of Conjunctival Hyperemia and Conjunctival Discharge Up to Day 6
Description: Percentage of patients that achieved clinical success, defined as achievement of a score of zero for both conjunctival hyperemia and conjunctival discharge in the study eye up to Day 6. Conjunctival hyperemia and conjunctival discharge were each assessed on a 4-point severity grade scale (0=none, +1=mild, +2=moderate, +3=severe).
Time Frame: 6 Days
Population: as for outcome 2
Measure: Number; unit: Percentage of Patients
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Number analyzed (Participants) | 166 | 167
Percentage of Patients | 51.8 | 41.3

ADVERSE EVENTS:
Description: Safety Population used for serious adverse event and adverse event analysis - defined as all patients who were randomized AND treated.
Arm/Group | Gatifloxacin 0.5% Eye Drops | Placebo Eye Drops
Serious Adverse Events (participants affected / at risk) | 2/429 | 0/427
Other Adverse Events (participants affected / at risk) | 19/429 | 26/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gatifloxacin 0.5% Eye Drops (N=429) | Placebo Eye Drops (N=427)
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gatifloxacin 0.5% Eye Drops (N=429) | Placebo Eye Drops (N=427)
Eye Irritation (Eye disorders) | 14 | 7
Conjunctivitis bacterial (Infections and infestations) | 5 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.